CLINICAL TRIAL: NCT06436898
Title: Proof of Concept of Hybrid Robotics for Gait Rehabilitation of Persons Post-stroke (PoCH-Rehab)
Brief Title: Proof of Concept of Hybrid Robotics for Gait Rehabilitation of Persons Post-stroke
Acronym: PoCH-Rehab
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Istituto Italiano di Tecnologia (Other); Istituto Nazionale di Ricovero e Cura per Anziani (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PoCH-Rehab
Record Dates: First submitted 2024-02-16; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Stroke Sequelae; Gait, Hemiplegic
Keywords: Gait rehabilitation; Exoskeleton; Functional Electrical Stimulation; Hemiplegia; Overground
MeSH Terms: conditions — Gait Disorders, Neurologic; Hemiplegia

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Assessor blind to treatment arm
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exoskeleton plus FES (Experimental): Participants will train gait with an overground exoskeleton and a combined myoelectrically controlled Functional Electrostimulation System (FES) applied to lower limb muscles during execution of gait.
  Interventions: Device: Combined overground gait exoskeleton and FES applied to lower limb
- Exoskeleton (Active Comparator): Participants will train gait with an overground exoskeleton.
  Interventions: Device: Overground gait exoskeleton

INTERVENTIONS:
Device: Combined overground gait exoskeleton and FES applied to lower limb — Gait rehabilitation for persons with stroke, with an overground exoskeleton combined with an electromyographically controlled FES applied to lower limb muscles during gait.
  Other Names: TWIN_Acta and FITFES
  Arms: Exoskeleton plus FES
Device: Overground gait exoskeleton — Gait rehabilitation for persons with stroke, with an overground exoskeleton.
  Other Names: TWIN_Acta
  Arms: Exoskeleton

SUMMARY:
Persons post-stroke suffer from hemiparesis affecting the functional abilities of the controlesional lower limb. Improving walking is therefore a primary rehabilitation goal for such patients. Robotic-Assisted Rehabilitation (RAR, e.g. exoskeletons) and Functional Electrical Stimulation (FES) are promising techniques to facilitate the functional recovery after stroke. allowing benefits to be maintained over long term.

DETAILED DESCRIPTION:
Exoskeletons were originally developed for subjects with spinal cord injury where they demonstrated a positive impact on rehabilitation and relative costs. The investigators expect the same trend also for stroke. Based on prior exploratory activities using an overgorund exoskeleton (TWIN_Acta) in gait rehabilitation post stroke, in this project the aim is to merge the potential of an overground exoskeleton and FES to treat the lower limb motor deficits in persons post-stroke, strengthening their residual abilities. Synchronized pairing of the two devices might boost the functional recovery of gait post-stroke by promoting neural reorganization The persons post stroke will undergo 20 gait rehabiliation sessions with the exoskeleton and with FES applied to the lower limb muscles during execution of gait with the aim of improving various gait and quality of life parameters. This experimental intervention will be compared to a control intervention using an exoskeleton alone for gait rehabiltation post stroke.

ELIGIBILITY:
Inclusion Criteria:

18 years or older

* Diagnosis of first unilateral ischemic or hemorrhagic ictus, at least two weeks from the event, ischemic or hemorrhagic
* diagnosis confermed with Computer Tomography or Magnetic Resonance Imaging
* 1 ≤ FAC (Functional ambulation category) ≤ 3
* 50 kg ≤ weight ≤ 90 kg
* 150 cm ≤ height ≤ 192 cm
* Femor length: 355-475 mm
* Tibia length: 405-485 mm
* Pelvic width 690-990 mm
* shoe size 36-45
* Capable of standing unsupported for at least one minute

Exclusion Criteria:

* Mini Mental State Examination score (corrected for age and education) < 24
* Clinical evidence in the medical records of visuospatial and ideomotor apraxia, behavioral disorders, neglect, severe visual and auditory sensory disorders or those which prevent use of the device
* patients at risk of fractures or with strategic fractures (unstabilized fractures or spinal instability)
* Major head trauma
* Subarachnoid hemorrhage, cerebral thrombosis
* Cardio-respiratory or internal clinical instability
* Pregnant or breastfeeding status;
* Recent malignant neoplasm
* Chronic inflammatory diseases with joint involvement of the lower limbs;
* Severe spasticity (Ashworth>3)
* Significant limitations in passive ROM of the hips and knees
* Problems with the integrity of the skin at the interface surfaces with the device or which would prevent sitting.
* Implanted electronic devices
* Epilepsy
* Severe peripheral neuropathies

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
System Usability scale (SUS) | At baseline and at post after 4 weeks of intervention
  The SUS assesses Usability and Acceptability of a device. The SUS consists of a 10 item questionnaire with five response options for respondents; from Strongly agree to Strongly disagree. The scores will be normalized to produce a percentile ranking. The higher the percentage the better the tested device is considiered.
Velocity of gait | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  Gait velocity during 3D gait analysis measured while walking overground over 10 meters. Velocity is measured in meters/second

SECONDARY OUTCOMES:
Motricity Index Lower limb (MI LL) | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  The motricity index is an ordinal method fo measuring limb strength. Maximum total lower limb score is 99. Scoring goes from 0 no movement to 33 normal power.
Fugl Meyer Assessment of motor recovery after stroke. Lower limb (FMA LL) | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  The scale evaluates and measures neuromotor recovery in post stroke patients. Items are scored on a 3-point ordinal scale, from 0 cannot perform to score 2 performs fully. Maximum score for lower limb is 34.
Functional Ambulation Category (FAC) | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  The FAC assesses functional ambulation in patients undergoing physical therapy. The clinician ticks a box of 5 broad categories of walking ability from not being able to walk or needing help from to or more persons to score of 5 if they can walk independently anywhere.
Stroke Rehabilitation Motivation Scale (7-item SRMS) | At baseline and at post after 4 weeks of intervention
  The 7-item SRMS was devised from the 28-item SRMS and inquires upon intrinsic and extrinsic motivation domains for rehabilitation. Scores range from 1 to 7 so the total score can range from 7-35 with higher scores indicating higher motivation.
Fatigue Severity Scale (FSS) | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  The impact of fatigue on day-to-day function is measured using the Fatigue Severity Scale (FSS). This measure is a self-report scale with nine questions answered on a 7-point Likert scale. The FSS score is reported as one total score which is the mean of the nine items. Scores range from 1 to 7 and higher scores indicate greater impact of fatigue on daily life.
Ashworth scale | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  The Modified Ashworth Scale (MAS) is a revised version of the original Ashworth Scale that measures spasticity in patients with lesions to the central nervous system. MAS is an assessment that is used to measure the increase in muscle tone. MAS assigns a grade of spasticity from a 0-4 ordinal scale with higher score indicating more spasticity. The grade is assigned by moving a joint/muscle through a high velocity quick stretch.Spasticity of calf and knee muscles will be tested
Manual muscle test (MMT) | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  MMT is a standardized set of assessments that measure muscle strength and function. Score range 0-5, minimum 0, maximum 5/5 meaning normal strength. Strength of calf and knee muscles will be tested.
Five times sit to stand test (5TStS) | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  The Five Times Sit to Stand Test measures one aspect of transfer skill. The test provides a method to quantify functional lower extremity strength and/or identify movement strategies a patient uses to complete transitional movements. Patient is timed while standing up and sitting down 5 times in row.
Timed up and go test (TUG) | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  The Timed Up and Go Test (TUG) assesses mobility, balance, walking ability, and fall risk. Patient are timed while standing up from a chair walking 3 meters, turning around, walking 3 meters and sitting down again.
  The patient sits in the chair with his/her back against the chair back. On the command "go," the patient rises from the chair, walks 3 meters at a comfortable and safe pace, turns, walks back to the chair and sits down.
  Timing begins at the instruction "go" and stops when the patient is seated.
Two minutes walking test (2MWT) | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  Walking capcaity is measured with the Participant timed while walking a 30 meter track constantly for 2 minutes. Participants are permitted to use their walking aids if necessary. The distance walked in 2 minutes is recorded and reported in metres
10 meter walking test (10MVT) | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  Walking speed is measured by the timed 10 m Walk Test (10MWT). Participants walk a distance of 10 m at their usual speed with their usual walking aids. Participants are timed while walking 10 meters from a starting point to an end point. Time taken from meter 2 to meter 8. Two repetitions are completed and the average time is used to calcualte walking speed in metres/second.
The walking handicap scale (WHS) | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  The walking handicap scale is a questionnaire asking subjective gait skills. The scale goes from 1 to 6, with score 1 being a physiological gait only with a physiotherapist, to score 6 being unrestricted community ambulation gait.
Beck Depression Inventory-II (BDI-II) | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  the BDI-II is a patient reported outcome that quantifies severity of depression. BDI-II identifies overt behavioral characteristics of depression. Items are on a four-point scale that ranges from 0 to 3. Ratings are summed to provide a total score ranging from 0 - 63. Scores >10 generally meet the threshold for a diagnosis of depression.
Unified Theory of Acceptance and Use of Technology (UTAUT) | At baseline and at post after 4 weeks of intervention
  A questionnaire asking how acceptable and easy to use the technological device is. The theoretical model of UTAUT suggests that the actual use of technology is determined by behavioural intention. The perceived likelihood of adopting the technology is dependent on the direct effect of four key constructs, namely performance expectancy, effort expectancy, social influence, and facilitating conditions. The UTAUT examines the acceptance of technology, determined by the effects of performance expectancy, effort expectancy, social influence and facilitating conditions.
Report of adverse events | at baseline and at post after 4 weeks of intervention
  Organized reporting of adverse events occurring during the use of the device
Euro Quality of Life-5 -dimension Questionnaire (EQ-5D-5L) | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  EQ-5D-FL is a standardized instrument for use as a measure of health for clinical and economic appraisal.Applicable to a wide range of health conditions and treatments, the EQ-5D health questionnaire provides a simple descriptive profile and a single index value for health status.
  Measures the 5 dimensions of:
  1. mobility
  2. self-care
  3. usual activities
  4. pain/discomfort
  5. anxiety/depression Each dimension is scored on a Likert scale of 5 levels, with higher scores indicating more severe problems.
Motion parameters derived from the kinematics of the body | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  Lower limb data will be captured utilizing two wearable Inertia Measurement Units (IMUs) operating at 280 Hz. These IMUs will be placed on both feet to analyze spatio-temporal gait characteristics. Through data processing, deviations from typical movement patterns will be quantified.
Postural capabilities will be evaluated based on body kinetics | At baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  Postural data of the lower limb will be acquired using an optoelectronic system combined with two force plates, sampling at 2000 Hz. Utilizing data processing techniques, deviations from normal postural dynamics will be determined.
Muscular synergies | at baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  Muscle synergies will be extracted from the Electromyography (EMG) envelope of each participant detected during overground gait employing the Non-Negative Matrix Factorization algorithm. Treatment-induced changes in the resemblance of muscle synergies to physiological patterns will be assessed. Module similarity will be gauged through the maximum scalar product of muscle weightings between each participant and the normative reference. Additionally, the activation profile similarity will be measured using the Pearson's correlation coefficient of each module's activation profile.
Instrumented 2 Minute Walk test (I2MWT) | at baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  Changes in the I2MWT will be evaluated through IMU sampling at 280 Hz positioned on the lower back. Deviations from the typical performance observed in healthy subjects will be evaluated.
Instrumented Timed Up and Go (ITUG) | at baseline, at post after 4 weeks of intervention, at follow up after 8 weeks from the end of intervention
  Changes in the instrumented Timed Up and Go (ITUG) test will be examined. The TUG test will be administered with an IMU sampling at 280 Hz positioned on the lower back. Deviations from the typical performance observed in healthy subjects will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Maurizio Ferrarin, PhD, Principal Investigator — Research Head of Biomedical Technology Department; Andrea Corsonello, PhD, Study Director — Research Head of the Neurological Unit
Locations (1):
- Fondazione Don Carlo Gnocchi IRCCS, Milan, Italy

IPD SHARING:
Plan to Share IPD: Yes
Data will be available upon request
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Preliminary data will be available at the end of the study February 2025
Access Criteria: at request to the Principal investigator